CLINICAL TRIAL: NCT00553605
Title: A Double-Blind, Double-Dummy, Randomized, Multicenter Study Comparing The Analgesic Efficacy And Safety Of Parecoxib 40mg I.V. To Ketoprofen 100mg I.V. In Renal Colic
Brief Title: Efficacy And Safety Of Parecoxib 40mg vs. Ketoprofen 100mg In The Management Of Acute Renal Colic
Acronym: NAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3481065
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2012-12

CONDITIONS: Pain
Keywords: Renal Colic Pain Urinary Tract Colic
MeSH Terms: conditions — Pain | interventions — Ketoprofen; parecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): Ketoprofen plus placebo parecoxib
  Interventions: Drug: Ketoprofen 100mg
- II (Active Comparator): Parecoxib plus placebo ketoprofen
  Interventions: Drug: Parecoxib 40mg

INTERVENTIONS:
Drug: Ketoprofen 100mg — Ketoprofen 100 mg diluted in 100 ml of normal sodium chloride solution into the established patient's IV line by slow injection in a 20-minute period; and IV dose of 2 ml of normal sodium chloride solution as placebo for Parecoxib by bolus injection
  Arms: I
Drug: Parecoxib 40mg — Parecoxib 40 mg diluted in 2 ml of normal sodium chloride solution administered by bolus injection; and an IV dose of 100 ml of normal sodium chloride solution as placebo for ketoprofen administered in a in a 20-minute period
  Arms: II

SUMMARY:
This is a multicenter, randomized, double blind, double dummy, comparative, active-controlled trial designed to assess the analgesic activity and safety of intravenous doses of parecoxib 40 mg relative to intravenous doses of ketoprofen 100 mg for the treatment of renal colic in outpatients presenting at emergency room settings. This trial is designed to show non-inferiority of parecoxib related to ketoprofen.

ELIGIBILITY:
Inclusion Criteria:

* Patient male or female with a confirmed diagnosis of acute renal colic with moderate to severe pain according to the VAS and Categoric pain scales

Exclusion Criteria:

* The patient has significant renal or hepatic conditions other than uncomplicated kidney stones.
* The patient has a history of clinically significant hypersensitivity to any NSAIDs, cyclooxygenase inhibitors, analgesics or sulfa medications which has a cross sensitivity to the medications used in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Brazil (6):
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Ribeirão Preto, São Paulo
  - Pfizer Investigational Site, São Bernardo do Campo, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
  - Pfizer Investigational Site, Vila Mariana - São Paulo, São Paulo
- Pfizer Investigational Site, Providencia, Santiago, RM, Chile
- Costa Rica (3):
  - Pfizer Investigational Site, Alajuela, Alajuela Province
  - Pfizer Investigational Site, Desamparados, Provincia de San José
  - Pfizer Investigational Site, San José, Provincia de San José
- Pfizer Investigational Site, Quito, Pichincha, Ecuador
- Pfizer Investigational Site, San Pedro Sula, San Pedro Sula, Honduras
- Pfizer Investigational Site, Lima, Lima Province, Peru

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3481065&StudyName=Efficacy%20And%20Safety%20Of%20Parecoxib%2040mg%20vs.%20Ketoprofen%20100mg%20In%20The%20Management%20Of%20Acute%20Renal%20Colic

RESULTS

PARTICIPANT FLOW:
Groups:
- Parecoxib: Single dose of parecoxib 40 milligram (mg) solution intravenously by bolus injection followed by single dose of 100 milliliter (mL) solution of placebo matched to ketoprofen intravenously by slow injection over 20 minutes.
- Ketoprofen: Single bolus injection of 2 mL solution of placebo matched to parecoxib followed by single dose of ketoprofen 100 mg solution intravenously by slow injection over 20 minutes.
Period: Overall Study
Arm/Group | Parecoxib | Ketoprofen
Started | 176 | 164
Treated | 174 | 164
Completed | 172 | 161
Not Completed | 4 | 3
Not completed — Did not meet entrance criteria | 1 | 3
Not completed — Did not receive full dose | 1 | 0
Not completed — Randomized but not treated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parecoxib | Ketoprofen | Total
Number analyzed (Participants) | 174 | 164 | 338
Age, Customized [Number; unit: participants]
  Less than (<) 18 years | 1 | 0 | 1
  18 to 44 years | 131 | 109 | 240
  45 to 64 years | 41 | 54 | 95
  Greater than or equal to (>=) 65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 61 | 125
  Male | 110 | 103 | 213

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Intensity Difference at 30 Minutes (mPID30min)
Description: mPID score was obtained by summation of product of length of the interval and difference in pain intensity (PI) divided by summation of length of the interval. Summation was done from zero to 30 minutes. Difference in pain intensity was obtained by subtracting the Pain Intensity Visual Analogue Scale (PI-VAS) at Minute 30 from baseline PI-VAS score. PI-VAS assessed with response to the question "How much pain are you having right now?" on a 100 millimeter (mm) line, with 0 mm=no pain, 100 mm= worst possible pain. mPID score ranged from -100 to 100. Positive score= improved response in pain.
Time Frame: Minute 30
Population: Per-protocol (PP): all randomized participants who received at least 1 dose of study drug; had 1 post-baseline pain assessment; no major protocol violations; received appropriate dose of study drug; had valid baseline, 15 and 30 min VAS pain assessments; did not take rescue medications for 30 min; had confirmed diagnosis of nephrolithiasis.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 156 | 141
mm | 34.147 (3.35) | 35.266 (3.46)
Statistical Analysis 1: Comparison: Parecoxib vs Ketoprofen; LS mean difference and 95 percent (%) confidence interval (CI) were based on analysis of covariance (ANCOVA) model with terms for treatment group and country, and baseline as covariates; Test type: Non-Inferiority or Equivalence — Non-inferiority was declared if the lower bound of the 2-sided 95% CI of the treatment difference (parecoxib - ketoprofen) was greater than -10 mm; Least-squares (LS) mean difference = -1.12, 95% CI 2-sided [-6.53 to 4.30], Standard Error of Mean 2.75

2. Secondary Outcome: Mean Pain Intensity Difference at 120 Min (mPID120min)
Description: mPID score was obtained by summation of product of length of the interval and difference in pain intensity (PI) divided by summation of length of the interval. Summation was done from zero to 120 minutes. Difference in pain intensity was obtained by subtracting the Pain Intensity Visual Analogue Scale (PI-VAS) at Minute 120 from baseline PI-VAS score. PI-VAS assessed with response to the question "How much pain are you having right now?" on a 100 millimeter (mm) line, with 0 mm=no pain, 100 mm= worst possible pain. mPID score ranged from -100 to 100. Positive score= improved response in pain.
Time Frame: Minute 120
Population: Modified intent- to-treat (mITT) included all randomized participants who received at least 1 dose of the study drug with at least 1 post-baseline pain assessment.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 173 | 164
mm | 51.608 (2.02) | 51.697 (2.05)
Statistical Analysis 1: Comparison: Parecoxib vs Ketoprofen; p-value, LS mean difference and 95% CI were based on ANCOVA model with terms for treatment group and country, and baseline as covariates; Test type: Superiority or Other; p = 0.972, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-5.04 to 4.86], Standard Error of Mean 2.52

3. Secondary Outcome: Time-specific Pain Intensity (PI) VAS Score
Description: PI-VAS assessed with response to the question "How much pain are you having right now?" on a 100 mm line, with 0 mm=no pain, 100 mm= worst possible pain.
Time Frame: Baseline, Minute 15, 30, 45, 60, 90, 120
Population: mITT included all randomized participants who received at least 1 dose of the study drug with at least 1 post-baseline pain assessment. Here 'n' signifies participants who were evaluable at specific time point for each treatment arm respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 173 | 164
mm
  Baseline (n= 173, 164) | 77.14 (17.92) | 76.99 (18.26)
  Minute 15 (n= 173, 164) | 50.42 (26.92) | 50.95 (24.65)
  Minute 30 (n= 172, 162) | 34.13 (28.57) | 33.65 (26.64)
  Minute 45 (n= 163, 156) | 21.75 (24.89) | 23.15 (24.93)
  Minute 60 (n= 156, 152) | 14.62 (21.25) | 17.53 (23.17)
  Minute 90 (n= 151, 144) | 9.80 (17.16) | 12.27 (20.22)
  Minute 120 (n= 147, 139) | 7.68 (14.29) | 8.02 (15.26)

4. Secondary Outcome: Time-specific Pain Intensity Difference (PID) at Minute 15, 30, 45, 60, 90 and 120
Description: PID score was obtained by subtracting the PI-VAS at each time point from baseline PI score. PI-VAS assessed with response to the question "How much pain are you having right now?" on a 100 mm line, with 0 mm=no pain, 100 mm= worst possible pain. PID score ranged from -100 to 100. Positive score= improved response in pain.
Time Frame: Baseline, Minute 15, 30, 45, 60, 90, 120
Population: mITT included all randomized participants who received at least 1 dose of the study drug with at least 1 post-baseline pain assessment. Here 'n' signifies participants who were evaluable at specific time points for each treatment arm respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 173 | 164
mm
  Minute 15 (n= 173, 164) | 26.72 (24.59) | 26.04 (26.13)
  Minute 30 (n= 172, 162) | 42.89 (28.70) | 43.22 (29.39)
  Minute 45 (n= 163, 156) | 54.37 (27.82) | 53.55 (27.98)
  Minute 60 (n= 156, 152) | 61.35 (25.44) | 59.34 (26.28)
  Minute 90 ( n= 151, 144) | 65.99 (22.88) | 64.33 (25.05)
  Minute 120 (n= 147, 139) | 68.07 (21.14) | 68.51 (21.21)
Statistical Analysis 1: Comparison: Parecoxib vs Ketoprofen; Minute 15: p-value, LS mean difference and 95% CI were based on ANCOVA model with terms for treatment group and country, and baseline as covariates; Test type: Superiority or Other; p = 0.768, ANCOVA; LS mean difference = 0.75, 95% CI 2-sided [-4.28 to 5.79], Standard Error of Mean 2.56
Statistical Analysis 2: Comparison: Parecoxib vs Ketoprofen; Minute 30: p-value, LS mean difference and 95% CI were based on ANCOVA model with terms for treatment group and country, and baseline as covariates; Test type: Superiority or Other; p = 0.866, ANCOVA; LS mean difference = -0.49, 95% CI 2-sided [-6.22 to 5.24], Standard Error of Mean 2.91
Statistical Analysis 3: Comparison: Parecoxib vs Ketoprofen; Minute 45: p-value, LS mean difference and 95% CI were based on ANCOVA model with terms for treatment group and country, and baseline as covariates; Test type: Superiority or Other; p = 0.729, ANCOVA; LS mean difference = 0.94, 95% CI 2-sided [-4.38 to 6.26], Standard Error of Mean 2.70
Statistical Analysis 4: Comparison: Parecoxib vs Ketoprofen; Minute 60: p-value, LS mean difference and 95% CI were based on ANCOVA model with terms for treatment group and country, and baseline as covariates; Test type: Superiority or Other; p = 0.290, ANCOVA; LS mean difference = 2.62, 95% CI 2-sided [-2.24 to 7.48], Standard Error of Mean 2.47
Statistical Analysis 5: Comparison: Parecoxib vs Ketoprofen; Minute 90: p-value, LS mean difference and 95% CI were based on ANCOVA model with terms for treatment group and country, and baseline as covariates; Test type: Superiority or Other; p = 0.314, ANCOVA; LS mean difference = 2.16, 95% CI 2-sided [-2.05 to 6.37], Standard Error of Mean 2.14
Statistical Analysis 6: Comparison: Parecoxib vs Ketoprofen; Minute 120: p-value, LS mean difference and 95% CI were based on ANCOVA model with terms for treatment group and country, and baseline as covariates; Test type: Superiority or Other; p = 0.926, ANCOVA; LS mean difference = 0.16, 95% CI 2-sided [-3.23 to 3.55], Standard Error of Mean 1.72

5. Secondary Outcome: Time-weighted Sum of Pain Relief Score Over 120 Min (TOTPAR120min)
Description: TOTPAR: time-weighted sum of Pain Relief (PR) over 120 min. TOTPAR score range was 0 (worst) to 480 (best). PR was assessed on a 5-point categorical pain relief rating scale wherein 0=No relief to 4=Complete relief.
Time Frame: Baseline through Minute 120
Population: mITT included all randomized participants who received at least 1 dose of the study drug with at least 1 post-baseline pain assessment. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 171 | 162
units on a scale | 362.42 (10.65) | 352.29 (10.85)
Statistical Analysis 1: Comparison: Parecoxib vs Ketoprofen; p-value, LS mean difference and 95% CI were based on ANCOVA model with terms for treatment group and country as covariates; Test type: Superiority or Other; p = 0.451, ANCOVA; LS mean difference = 10.13, 95% CI 2-sided [-16.3 to 36.54], Standard Error of Mean 13.43

6. Secondary Outcome: Number of Participants With Pain Relief (PR)
Description: PR was assessed on a 5-point categorical pain relief rating scale wherein 0= None, 1= a little, 2= Some, 3= a lot and 4= Complete relief.
Time Frame: Minute 30, 120
Population: mITT included all randomized participants who received at least 1 dose of the study drug with at least 1 post-baseline pain assessment. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this measure and 'n' signifies participants who were evaluable at specific time point for each treatment arm respectively.
Measure: Number; unit: participants
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 171 | 162
participants
  Minute 30: none (n= 171, 162) | 10 | 9
  Minute 30: a little (n= 171, 162) | 21 | 19
  Minute 30: some (n= 171, 162) | 35 | 44
  Minute 30: a lot (n= 171, 162) | 74 | 65
  Minute 30: complete (n= 171, 162) | 31 | 25
  Minute 120: none (n= 146, 139) | 1 | 1
  Minute 120: a little (n= 146, 139) | 0 | 4
  Minute 120: some (n= 146, 139) | 16 | 8
  Minute 120: a lot (n= 146, 139) | 40 | 46
  Minute 120: complete (n= 146, 139) | 89 | 80
Statistical Analysis 1: Comparison: Parecoxib vs Ketoprofen; Minute 30: p-value was calculated using Cochran-Mantel-Haenszel (CMH) model and using modified ridit scores, testing for non-zero correlation and controlling for country; Test type: Superiority or Other; p = 0.3982, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Parecoxib vs Ketoprofen; Minute 120: p-value was calculated using Cochran-Mantel-Haenszel (CMH) model and using modified ridit scores, testing for non-zero correlation and controlling for country; Test type: Superiority or Other; p = 0.5552, Cochran-Mantel-Haenszel

7. Secondary Outcome: Number of Participants With Response in Pain Intensity
Description: PI-VAS assessed with response to the question "How much pain are you having right now?" on a 100 mm line, with 0 mm=no pain, 100 mm= worst possible pain. Responders were those who had a decreased in VAS of at least 20 mm.
Time Frame: Minute 30
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 172 | 162
participants | 132 | 124
Statistical Analysis 1: Comparison: Parecoxib vs Ketoprofen; p-value was based on logistic regression model with terms for treatment group and baseline as covariates; Test type: Superiority or Other; p = 0.9785, Regression, Logistic; Odds Ratio (OR) = 1.007, 95% CI 2-sided [0.60 to 1.69]

8. Secondary Outcome: Patient's Global Evaluation of Study Medication
Description: Participants' response to the question "How would you rate the study medication you received for pain?" on a 4-point categorical scale, 1=Poor, 2= Fair, 3=Good, 4=Excellent was evaluated.
Time Frame: Minute 30, 120
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 172 | 163
participants
  Minute 30: poor | 12 | 10
  Minute 30: fair | 21 | 17
  Minute 30: good | 76 | 66
  Minute 30: excellent | 63 | 70
  Minute 120: poor | 8 | 5
  Minute 120: fair | 16 | 16
  Minute 120: good | 49 | 46
  Minute 120: excellent | 98 | 96
Statistical Analysis 1: Comparison: Parecoxib vs Ketoprofen; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.2482, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Parecoxib vs Ketoprofen; Minute 120: p-value was calculated using CMH model and using modified ridit scores, testing for non-zero correlation and controlling for country; Test type: Superiority or Other; p = 0.7659, Cochran-Mantel-Haenszel

9. Secondary Outcome: Physician's Global Evaluation of Study Medication
Description: Physicians' response to the question "How would you rate the study medication the patient received for pain?" on a 4-point categorical scale, 1=Poor, 2= Fair, 3=Good, 4=Excellent was evaluated.
Time Frame: Minute 30, 120
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 172 | 163
participants
  Minute 30: poor | 11 | 11
  Minute 30: fair | 22 | 23
  Minute 30: good | 69 | 63
  Minute 30: excellent | 70 | 66
  Minute 120: poor | 8 | 8
  Minute 120: fair | 14 | 15
  Minute 120: good | 45 | 45
  Minute 120: excellent | 104 | 95
Statistical Analysis 1: Comparison: Parecoxib vs Ketoprofen; Minute 30: p-value was calculated using CMH model and using modified ridit scores, testing for non-zero correlation and controlling for country; Test type: Superiority or Other; p = 0.9783, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Parecoxib vs Ketoprofen; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.6847, Cochran-Mantel-Haenszel

10. Secondary Outcome: Number of Participants With Use of Rescue Medication (RM)
Description: Rescue medications included intravenous 0.1 to 0.2 mg/kilogram (kg) of morphine or 1 mg/kg of pethidine or muscle relaxants.
Time Frame: Up to Minute 120
Population: mITT included all randomized participants who received at least 1 dose of the study drug with at least 1 post-baseline pain assessment.
Measure: Number; unit: participants
Arm/Group | Parecoxib | Ketoprofen
Number analyzed (Participants) | 173 | 164
participants | 26 | 25
Statistical Analysis 1: Comparison: Parecoxib vs Ketoprofen; Test type: Superiority or Other; p = 0.9645, Log Rank

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Parecoxib | Ketoprofen
Serious Adverse Events (participants affected / at risk) | 9/174 | 8/164
Other Adverse Events (participants affected / at risk) | 47/174 | 55/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parecoxib (N=174) | Ketoprofen (N=164)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Condition aggravated (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 2 | 7
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parecoxib (N=174) | Ketoprofen (N=164)
Bradycardia (Cardiac disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 7 | 5
Vomiting (Gastrointestinal disorders) | 4 | 5
Chills (General disorders) | 1 | 2
Pain (General disorders) | 6 | 9
Pyrexia (General disorders) | 3 | 1
Vessel puncture site pain (General disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 7 | 2
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 4
Paraesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 3 | 0
Renal pain (Renal and urinary disorders) | 0 | 1
Urethral pain (Renal and urinary disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Angiopathy (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
PR at all time points, proportion of participants with >= 1 grade improvement in PR 30 min were replaced by PR at 30 and 120 min; number of participants with response in PI included; time to RM reported as number, due to change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.